CLINICAL TRIAL: NCT04635800
Title: A First-in-human, Open-label, Single Ascending Dose Study to Assess Safety and Tolerability of Intravitreal MHU650 in Participants With Macular Edema From Diabetic Macular Edema (DME), Neovascular Age-related Macular Degeneration (nAMD), or Retinal Vein Occlusion (RVO)
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of IVT MHU650 in Macular Edema Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMHU650A12101
Record Dates: First submitted 2020-11-13; First posted 2020-11-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Macular Edema; Diabetic Macular Edema; Neovascular Age-related Macular Degeneration; Retinal Vein Occlusion
Keywords: Macular degeneration; age-related macular degeneration; dry macular degeneration; wet macular degeneration; Diabetic Macular Edema; DME; Neovascular age-related macular edema; nAMD; Retinal Vein Occlusion; RVO; MHU650; macular edema
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion; Macular Degeneration; Geographic Atrophy; Wet Macular Degeneration

STUDY DESIGN:
Intervention Model Description: The primary objective of this open-label study is to evaluate the initial safety, tolerability, and pharmacokinetics (PK) of single IVT doses of MHU650 in up to 24 patients. The screening period will be up to 60 days. A single dose of MHU650 will be administered at Baseline / Day 1 in the study eye. The follow up period will last until Day 60 / end of study (EOS). A post study safety phone contact call will occur 30 days after the EOS visit. A total of up to 4 cohorts may be enrolled, with an additional optional lower or intermediate cohort of 6 participants.
Masking Description: Open-label; no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Cohort 1; open-label, non-randomized, single administration
  Interventions: Drug: MHU650
- Cohort 2 (Experimental): Cohort 2; open-label, non-randomized, single administration
  Interventions: Drug: MHU650
- Cohort 3 (Experimental): Cohort 3, open-label; non-randomized, single administration
  Interventions: Drug: MHU650
- Cohort 4 (Experimental): Cohort 4, open-label, non-randomized, single administration
  Interventions: Drug: MHU650

INTERVENTIONS:
Drug: MHU650 — MHU650 powder for solution for injection

SUMMARY:
This was an open-label, multi-center, FIH study with a single ascending dose (SAD) design that assessed the safety, tolerability and pharmacokinetics (PK) of a single IVT dose of MHU650 in up to 24 participants with macular edema.

DETAILED DESCRIPTION:
A total of up to 4 cohorts were planned to be enrolled, with an additional lower or intermediate cohort of participants. First to third generation Japanese participants could be enrolled in all cohorts but were not required to be enrolled. The screening period for this study will be up to 60 days. A single dose of MHU650 intravitreal injection will be administered at Baseline / Day 1 in the study eye. The follow up period will last until Day 60 / end of study (EOS). A post study safety phone contact call will occur 30 days after the EOS visit.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with macular edema in at least one eye, including those with focal or diffuse diabetic macular edema (DME), neovascular age-related macular degeneration (nAMD), or retinal vein occlusion (RVO). In the opinion of the investigator, the decrease in vision in the study eye must be due to macular edema.
* Early Treatment Diabetic Retinopathy (ETDRS) letter score in the study eye must equal to or worse than 60 letters (approximately Snellen equivalent of 20/63) but better than 14 letters (20/500) at screening and baseline. The ETDRS score in the non-study eye should be ≥ 60 letters at screening and baseline.
* Sufficiently clear ocular media and adequate pupil dilation to permit fundus photographs of adequate clarity to measure diameters of retinal arteries and veins
* Vital signs as specified in the protocol

Key Exclusion Criteria:

* Concomitant conditions or ocular disorders in the study eye which may, in the opinion of the investigator, confound the interpretation of study results, compromise visual acuity or require medical or surgical intervention during the study period
* High risk and/or/ active proliferative diabetic retinopathy in the study eye, as per investigator assessment at both screening and baseline.
* Participants with the following conditions in the study eye at screening or baseline must be excluded: structural damage of the fovea, vitreous hemorrhage, retinal detachment, vitreomacular traction, macular hole, retinal arterial occlusion, neovascularization of iris of any cause.
* Laser photocoagulation (macular or panretinal) in the study eye during the 6-month period prior to baseline.
* Patients with type 1or type 2 diabetes who have hemoglobin A1C of ≥ 12 at screening
* Other ocular conditions as specified in the protocol
* Systemic conditions as specified in the protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with ocular and nonocular adverse events | Day 1 to Day 60
  An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Change from baseline in Best Correct Visual Acuity (BCVA ) by dose level and timepoint - Study Eye | Day 1 to Day 60
  Best Correct Visual Acuity was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
Change from baseline in Central subfield thickness (CSFT) (µm) in the study eye by dose level and timepoint | Day 1 to Day 60
  Central subfield thickness was measured by spectral domain optical coherence tomography (SD-OCT).
Change from baseline in Intraocular pressure (IOP) (mmHg) in the study eye by dose level and timepoint | Day 1 to Day 60
  Intraocular pressure was measured per the sites' local standard operating procedures, via tonometry.

SECONDARY OUTCOMES:
Pharmacokinetics of single dose of MHU650 - Cmax | Days 1, 2, 5, 15, 29, 43 and 60
  Assess serum PK profile of MHU650 by Cmax (if feasibile)
Pharmacokinetics of single dose of MHU650 - Tmax | Days 1, 2, 5, 15, 29, 43 and 60
  Assess serum PK profile of MHU650 by Tmax (if feasibile)
Pharmacokinetics of single dose of MHU650 - T1/2 | Days 1, 2, 5, 15, 29, 43 and 60
  Assess serum PK profile of MHU650 by T1/2 (if feasibile)
Pharmacokinetics of single dose of MHU650 - AUClast | Days 1, 2, 5, 15, 29, 43 and 60
  Assess serum PK profile of MHU650 by AUClast (if feasibile)
Pharmacokinetics of single dose of MHU650 - AUCinf | Days 1, 2, 5, 15, 29, 43 and 60
  Assess serum PK profile of MHU650 by AUCinf (if feasibile)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (5):
  - Novartis Investigative Site, Huntington Beach, California
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Hagerstown, Maryland
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Houston, Texas
- Novartis Investigative Site, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CMHU650A12101 from the Novartis Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18049
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1501